CLINICAL TRIAL: NCT02460848
Title: Effects of Unconditional Cash Transfers on the Management of Severe Acute Malnutrition (SAM) in the Democratic Republic of Congo: a Cluster Randomized Trial
Brief Title: Effects of Cash Transfers on Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNICEF (Other)
Collaborators: Save the Children (Other)
Responsible Party: Principal Investigator, Emmanuel Grellety, Principal Investigator, UNICEF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ARCCII-Nutrition
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Severe Malnutrition
Keywords: Malnutrition; Severe Acute Malnutrition; Cash Transfer; Democratic Republic of Congo; Cluster randomize trial
MeSH Terms: conditions — Malnutrition; Severe Acute Malnutrition | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outpatient therapeutic program, counseling and cash transfer (Experimental): Ten outpatient therapeutic program sites (OTP) will be randomly allocated to unconditional cash transfer for children admitted for treatment of SAM according to the integrated management of acute malnutrition national protocol which will be associated with counseling on infant and young child feeding (IYCF).
  Interventions: Other: Outpatient therapeutic program, counseling and cash transfer
- Outpatient therapeutic program and counseling (Active Comparator): Ten outpatient therapeutic program sites (OTP) will be randomly allocated for children admitted for treatment of SAM according to the integrated management of acute malnutrition national protocol which will be associated with counseling on infant and young child feeding (IYCF).
  Interventions: Other: Outpatient therapeutic program and counseling

INTERVENTIONS:
Other: Outpatient therapeutic program, counseling and cash transfer — Each household will receive an unconditional cash transfer of $40 value every month during a 6 months' period.
  The amount of cash per household per month was defined according to the results of the Household Economy Approach survey. This amount represents 70% of supplement to the monthly average household income characterized as very poor to meet their basic needs. This threshold corresponds to the total of food and income necessary to cover 100% of energy needs food (2100 kcal per day per person), the costs associated with the preparation and consumption of food (e.g. salt, soap, kerosene and / or firewood for cooking and basic lighting) and finally all expenses for access to water for human consumption.
  Arms: Outpatient therapeutic program, counseling and cash transfer
Other: Outpatient therapeutic program and counseling
  Arms: Outpatient therapeutic program and counseling

SUMMARY:
Cash transfer, aims to strengthen food security for vulnerable households by giving families enough purchasing power to consume an adequate and balanced diet, maintain a good standard of hygiene, access health services, and invest in their own means of food production in addition to their children's growth and development.

While cash transfer to vulnerable households has shown a long-term positive impact on growth and on malnutrition-related mortality in children aged 0-5 years, there is little conclusive evidence their effectiveness in Sub-Saharan Africa that cash transfer has a direct effect on the Community-based Management of Acute Malnutrition (CMAM). Here, the investigators will perform a cluster-randomized trial to investigate during 6 months the effects of unconditional cash transfers on the management of severe acute malnutrition (SAM) in children from 6 to 59 months according to the national protocol in the Democratic Republic of Congo.

ELIGIBILITY:
Inclusion Criteria:

* Living in the catchment area of one of the 20 outpatient therapeutic program site participating in this cluster randomized trial;
* 6-59 months of age;
* Weight for Height Zscore <-3 SD (WHO Growth Standards 2006) and/or Mid-Upper Arm Circumference <115mm and/or with bilateral edema;
* No major clinical complications;
* Positive appetite test;
* Accept to participate at the study.

Exclusion Criteria:

* Not living in the catchment area of the outpatient therapeutic program site of the cluster randomized trial;
* Weight-for-Height Z-score ≥-3 (WHO Growth Standards 2006) and Mid-Upper Arm Circumference ≥115mm without bilateral edema;
* Major clinical complications;
* Failure to appetite test;
* Refuse to participate at the study.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1600 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Recovery rate in the outpatient therapeutic program | At 6 week
  Recovery is defined for patient of 6 to 59 months old as Weight-for-Height Z-score ≥-1.5 SD (WHO Growth Standards 2006) or Mid-Upper Arm Circumference ≥125mm at two consecutive visits and absence of bilateral edema for 14 days.

SECONDARY OUTCOMES:
Recovery rate in the outpatient therapeutic program | At 8 week
Length of stay in the outpatient therapeutic program | One month (average)
Default rate in the outpatient therapeutic program | Two weeks
  Patient who failed to appear for two consecutive weeks during the follow-up visits.
Relapse rate | At 2, 3 and 4 months following discharge
  Patient who reach inclusion criteria within 2 months following discharge.
Transfer rate from outpatient therapeutic program to inpatient therapeutic program | One month average
  Patient who develop signs of a serious medical complication according to the national protocol are transfer to the inpatient therapeutic program.
Failure rate in the outpatient therapeutic program | Up to three months
  Patients who failed to reach after 3 months the recovery criteria.
Morbidity rate | At 6 week, 8 week and 6 month
  ARI, diarrhoea, anaemia and malaria incidence. Morbidity will be assessed every week in the outpatient therapeutic program and every month after discharge by a locally pre-tested standardized questionnaire.
Death rate | At 6 week, 8 week and 6 month
  Death from any cause during follow-up.
Weight gain | At 6 week, 8 week and 6 month
  Weight gain will be assessed every week in the outpatient therapeutic program and every month after discharge.
Mid-Upper Arm Circumference gain | At 6 week, 8 week and 6 month
  Mid-upper arm circumference gain will be assessed every week in the outpatient therapeutic program and every month after discharge.
Change in Growth rates | At 6 month
  Growth will be measured every week in the outpatient therapeutic program and every month after discharge.
Diet replacement & Intra-household dispatching of the therapeutic food | One month average
  Diet replacement & Intra-household dispatching of the therapeutic food will be assessed with the household every week during the recovery period by a locally pre-tested standardized questionnaire.
Change in the Individual Dietary Diversity Score (IDDS) | At 6 week, 8 week and 6 month
  IDDS for measurement of food access of the children will be assessed with the household every week during the recovery period and every month after discharge by a locally pre-tested standardized questionnaire.
Change in the Household Dietary Diversity Score (HDDS) | At 6 month
  HDDS for measurement of food access will be assessed with the household at the beginning and the end of the study by a locally pre-tested standardized questionnaire.
Satisfaction of parents and acceptability | At 6 month
  Survey will be conducted in the households at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Alain Ategbo, PhD, Study Chair — United Nations Children's Fund (UNICEF)
Locations (1):
- Save the Children, Mbuji-Mayi, East Kasai, Democratic Republic of the Congo

REFERENCES:
- [Derived] Grellety E, Babakazo P, Bangana A, Mwamba G, Lezama I, Zagre NM, Ategbo EA. Effects of unconditional cash transfers on the outcome of treatment for severe acute malnutrition (SAM): a cluster-randomised trial in the Democratic Republic of the Congo. BMC Med. 2017 Apr 26;15(1):87. doi: 10.1186/s12916-017-0848-y. PMID 28441944